CLINICAL TRIAL: NCT01321151
Title: Use of Resveratrol to Decrease Secondary Brain Injury Following Sports-Related Concussions: a Double-Blind, Placebo-Controlled Study
Brief Title: Use of Resveratrol to Decrease Acute Secondary Brain Injury Following Sports-Related Concussions in Boxers
Acronym: REPAIR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Joshua Gatson, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU 092010-188
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Sports Concussion
Keywords: Mild Brain Injury; Concussions; Resveratrol; Boxers; ImPACT; MRI
MeSH Terms: conditions — Tooth, Impacted | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo
- Resveratrol (Experimental): Intervention
  Interventions: Drug: Resveratrol

INTERVENTIONS:
Drug: Resveratrol — The dose of resveratrol is 500 mg. The route of administration is oral, once-a-day for 30 days after injury.
  Arms: Resveratrol
Drug: Placebo — The placebo is a sugar pill. The route of administration is oral, once-a-day for 30 days after injury.
  Arms: Sugar Pill

SUMMARY:
Sports-related concussions are a serious problem in football, boxing, and other full contact sports. After experiencing consecutive concussions, there is an increase in neurological deficits that can lead to long-term cognitive problems (Dementia pugilistica). To combat this increase in brain damage, novel strategies need to be developed to protect athletes that are participating in these full contact sports. The purpose of this study is to elucidate whether resveratrol decreases brain injury and improves brain function after experiencing a concussion in boxers.

DETAILED DESCRIPTION:
Each year, approximately 3 million sports-related concussions occur in athletes. Only about 5% of these concussions are treated in the hospital setting. To date, there are no effective interventions used at decreasing the levels of oxidant injury and inflammation within these athletes. The standard form of care in these athletes is usually rest and light exercise for 1 -2 weeks, before returning to the sport. Within this brain injury population, administration of a neuro-protectant agent immediately following the concussion may alleviate or prevent secondary injury and subsequent development of long-term cognitive deficits such as Chronic Traumatic Encephalopathy (CTE) and Dementia pugilistica (DP). Since sports-related concussions are a serious problem in our youth, by using safe interventions, we believe that the levels of oxidant injury and brain inflammation will be decreased. In addition, these neuro-protective agents may improve cognition in these boxers, and decrease the incidence of DP.

Following brain injury, the secondary injury that immediately follows consists of heightened damage by oxygen radicals, which in turn damages vital lipids, proteins, and nucleic acids. This damage is exacerbated by highly acidic conditions with lead to the release of iron and the production of more harmful oxygen radicals. An increase in these oxygen radicals has been observed from minutes to hours within the primary injury. In addition, there is an increase in inflammation as well as excitotoxicity in the brain after traumatic injury. To combat this secondary injury, the use of anti-oxidants in individuals is warranted to decrease the amount of brain damage and cognitive decline after experiencing a severe brain injury. For example, resveratrol (3,5,4'-trihydroxystilbene) which is a polyphenol compound that is commonly found in grapes, is a nutritional supplement with anti-oxidant and anti-inflammatory properties with great promise for treating TBI secondary injury. A number of researchers have demonstrated that resveratrol protect multiple organs (heart, kidney, brain) from ischemia after injury. With respect to the brain, resveratrol has been shown to protect from oxidative stress, Huntington's disease, and stroke. Additionally, following TBI in various animal models, resveratrol protected from severe brain injuries. Results from these brain studies suggest that resveratrol protects from a plethora of injuries and may afford protection from secondary injury in individuals suffering from a severe brain injury.

In this pilot clinical trial, boxers (n=30) will be consented to participate in this study prior to engaging in a boxing match. The concussion history will be collected before enrolling. Baseline cognitive testing and magnetic resonance imaging (MRI) scan will be performed to obtain both structural and functional data. Only 12 boxers that have a concussion will be enrolled in this study. After participating in the boxing match, if the boxer has been diagnosed with having a concussion by the ringside physician, the boxers will be treated with an oral dose of the active trans-resveratrol (500 mg) or placebo within 2 hours of completion of the boxing match. The boxer will be treated with either resveratrol or placebo (depending on the randomization schedule) once a day for 30 days. Cognitive testing and MRI scans will be conducted on day 7 after the concussion.

ELIGIBILITY:
Inclusion Criteria:

1. Boxers between the ages 18-35 years old
2. Both men and women
3. Boxers with an estimated concussion (Mild and Moderate) as estimated by the on-site physician or athletic trainer
4. Subject has provided full written informed consent prior to the performance of any protocol-specified procedure

Exclusion Criteria:

1. Immediate hospitalization for sports-related concussion (Severe Concussion)
2. Known inclusion in an interventional clinical trial
3. Patients with metal implants that would interfere with the MRI scan
4. Known anemia
5. Known Pregnancy
6. Known history of alcohol/drug abuse

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua W. Gatson, Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | Resveratrol
Started | 6 (The boxer was treated once-a-day for 30 days.) | 6 (The boxer was treated with once-a-day for 30 days.)
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Resveratrol | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5) | 27 (5.3) | 26 (5.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 0 | 2 | 2
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Liver Function Testing (Aspartate Transaminase [AST]/Alanine Transaminase [ALT] Ratios) to Screen for Adverse Events.
Description: Liver Function Tests will be conducted on day 7 after concussion.
Time Frame: Day 7 post concussion
Population: This Outcome measure differs from Outcome measure 1 based on the time frame. In Outcome measure 1, the time frame listed is -'30 Days post concussion' whereas within Outcome measure 2, the time frame listed is -'Day 7 post concussion'.
Measure: Mean (Standard Deviation); unit: AST/ALT ratio
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 6 | 6
AST/ALT ratio | 1.57 (.4) | 1.24 (.3)

2. Primary Outcome: Liver Function Testing (Aspartate Transaminase [AST]/Alanine Transaminase [ALT] Ratios) to Screen for Adverse Events.
Description: Liver Function Tests will be conducted on day 30 after concussion.
Time Frame: 30 Days post concussion
Population: No data was collected for30 days post concussion
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Functional Connectivity in Concussed Boxers
Description: Functional connectivity magnetic resonance imaging
Time Frame: 30 Days
Population: No data was collected for 30 days post concussion
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Reaction Time Composite as Assessed by Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) Cognitive Test Performance
Description: The reaction time composite score (range 0.5-0.8) is an average of: modules 3,4, 5, then divided by 3.The higher the composite score, the worse the outcomes.
  1. Average correct reaction time of interference stage of module 3 (X's and O'S) - Measures the number of correctly identified items (total possible correct =12), scoring 0-12. There is 4 trials of this module completed. Measures the average reaction time for correct responses on the interference (distracter) test
  2. Average correct reaction time of module 4 (Symbol Match) - Provides the number of correct matches out of 27 when the symbol number pairings are visible. The quicker the response time for each correctly identified symbol match indicates a better outcome.
  3. Average correct reaction time of module 5 (Color Match) - is number of correct color matches. The quicker the response time to a correct color match is a better outcome.
  Each modules is measured in percentage correct
Time Frame: 7 days post concussion
Measure: Mean (Standard Deviation); unit: Composite Score
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 6 | 6
Composite Score | .675 (.103) | .695 (.179)

5. Secondary Outcome: Reaction Time Composite as Assessed by Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) Cognitive Test Performance
Description: as for outcome 4
Time Frame: 24-72 hours post concussion
Population: No data was collected for 24-72 hours post concussion
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Reaction Time Composite as Assessed by Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) Cognitive Test Performance
Description: as for outcome 4
Time Frame: 30 days post concussion
Population: No data was collected for 30 days post concussion
Arm/Group | Sugar Pill | Resveratrol
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Resveratrol
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes